CLINICAL TRIAL: NCT04635930
Title: Effects of Taping Verses Traditional Exercises on Scapular Stabilization and Upper Limb Function in Hemiplegic Cerebral Palsy.
Brief Title: Taping and Traditional Exercises in Upper Limb Function in Hemiplegic
Acronym: CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00685 Mahnoor Ayaz
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taping plus Traditional exercises (Experimental): kinesio tape for improving the alignment of the scapula by inhibiting the hyperactive upper trapezius and facilitating the weak serratus anterior muscleStretching of the tight muscles of upper limb.
  * Reaching forward sidewise and backward.
  * Strengthening of the weak muscles by resisted exercise. 2-3 sets of 8-12 repetition, 4 times per week (ACSM guidelines).
  * Prone lying weight bearing on elbows (four point kneeling)
  * side sitting with weight bearing on the effected side, for 5 minutes.
  * Wall pushups.
  * Catching and throwing of ball
  Interventions: Other: Taping plus Traditional exercises
- Traditional exercises (Active Comparator): Stretching of the tight muscles of upper limb.
  * Reaching forward sidewise and backward.
  * Strengthening of the weak muscles by resisted exercise. 2-3 sets of 8-12 repetition, 4 times per week (ACSM guidelines).
  * Prone lying weight bearing on elbows (four point kneeling)
  * side sitting with weight bearing on the effected side, for 5 minutes.
  * Wall pushups.
  * Catching and throwing of ball
  Interventions: Other: Taping plus Traditional exercises

INTERVENTIONS:
Other: Taping plus Traditional exercises — The children will be taped 6 days per week for a total a period of 08 weeks. The tape will be used and keep the scapula in position for 3 days and the region will then be left to rest for 24 hours. Kinesio Taping will then be re-applied by the same experienced research assistants for another 3 days.

SUMMARY:
The aim of this research is to determine the Effects of taping verse traditional exercises on scapular stabilization and upper limb function in hemiplegic cerebral palsy.Taping and traditional exercises effects on scapular stabilization and support upper limb fuction in Hemiplegic cerebral palsy patients. A randomized controlled trial will be done at hayatabad Medical Complex Peshawar. The sample size is 26. The Participants will be divided into two groups, 13 participants in group A and 13 in Group B. The study duration will 6 months. Sampling technique will purposive non probability sampling technique. Only 6 to 8 years participants with Hemiplegic cerebral palsy will be included. Tools will be used in this study are Quality of upper extremity skill test, The Functional Independence Measure for Children (WeeFIM): Data will be analyzed through Statistical Package of Social Sciences version23.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a non-progressive group of developmental motor disorders that may result in spasticity, paralysis, or abnormal posture. Muscle weakness has been recognized as a primary clinical feature in CP. It is the most common cause of physical disability in children, with a prevalence of 2 to 2.5 per 1000 live births in Western countries . Hemiplegia is a form of spastic Cerebral Palsy (CP) in which one arm and leg on either the right or left side of the body is affected. There are several sub-types of CP, one of which is spastic hemiplegic CP, which occurs in approximately23%ofchildren with spastic CP. Because CP is a lifelong condition, all aspects of an individual's development and independence are impacted. The upper limb is usually more severely involved than lower one. This limits reaching, grasping and object manipulation, interfering also with exploration, play, self-care and other activities of daily living. Children with hemiplegic cerebral palsy often have marked hand involvement with excessive thumb adduction and ﬂexion and limited active wrist extension from infancy. Deficits in upper limb motor function can affect a 53 child's participation in self-care and play, and thus interfere with development in 54 multiple domains. Chronic hemiplegic patient with residual scapular weakness has the spasticity of some of the scapular muscles, which disturb the proximal stability of the scapulothoracic joint.This limits reaching, grasping and object manipulation, interfering also with exploration, play, self-care and other activities of daily living. Becoming independent in activities of daily living requires amongst others a smooth coordination between both hands

* Though motor deficits have been emphasized, sensory dysfunction may exist and may contribute to diminished use of the affected hand. Several studies have emphasized the impact that sensory deficits may have on hand function, because precise motor ability is dependent on sensory input. Common treatments include botulinum toxin, orthopedic surgery constraint induced movement therapy, pharmacotherapy for muscle tone, occupational therapy and traditional physiotherapy. As impairments in these children involve a variable range of functions, the children need comprehensive rehabilitation therapy
* A study conducted on ''Neuromuscular taping for the upper limb in Cerebral Palsy'' discussed that, the data showed that, after the intervention, the movement of the affected arm was faster, in particular in the adjusting and returning phase. The movement was also smoother and with a more physiological range of motion at shoulder and elbow. After the taping removal, Researcher found in fact a reduction of the adjusting and returning phase duration, a lower value of average jerk parameter and improved upper limb ranges of motion if compared to pre-test condition . A study on ''the effect of taping on scapular stability and upper limb function in recovering hemiplegics with scapular weakness'' shows that scapular taping has improved the functional outcome in upper extremity hemiplegics with scapular weakness. Scapular taping has improved the alignment of the scapula by inhibiting the hyperactive upper trapezius and facilitating the weak serratus anterior muscle by altering length-tension properties of muscles and providing kinesthetic awareness of scapular position during rest and movement of upper extremity. A study on Functional Impact of Shoulder Taping in the Hemiplegic Upper Extremity reported relief of pain symptoms immediately after being taped. Reduction in the patient's subjective sense of pain was associated with improvements in the ability to perform activities of daily living (ADL) and in range of motion (ROM). The patient showed improvements in the ability to dress, toilet, and bathe himself following shoulder taping and concomitant reduction in pain. The reported changes in ROM were less dramatic than the ADL improvement .A systematic review on the effects of elastic therapeutic taping on motor function in children with motor impairments. From the studies analyzed, it appears that interest in the use of elastic therapeutic taping as an adjunct and assistance resource to conventional treatment has grown over the last decade.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as hemiplegic cerebral palsy.
* Age group 7 to 14 years.
* Both males and females.
* Hemiplegic patients demonstrating weakness of scapular muscles i.e., less than grade 3 on manual muscle testing scale.

Hemiplegics who understand and follow verbal commands.

Exclusion Criteria:

* Hemiplegic patient with cognitive and perceptual disorders.

  * Hemiplegic patient having sensory, behavioral dysfunction and emotional liability.
  * Hemiplegic patient who is having any associated history of trauma and other medical disorders of hemiplegic upper extremity.
  * Any musculoskeletal structural disorder impeding upper limb function.
  * Participating in any experimental rehabilitation or drug studies.
  * Excessive spasticity that is score of >3 on modified Ashworth spasticity scale

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Quality of upper extremity skills test | 8 weeks
  The Quality of upper extremity skills test (QUEST) This measures the upper limb function in four domains, dissociated movements grasp of hand, weight bearing of upper limb and protective extension of upper limb including 33 items. Each item comprises, however, several sub items and both left and right upper extremity is assessed, so a total of 174. This is designed to be used with children who exhibit neuromotor dysfunction with spasticity and has been validated with children 18 months to 8 years.

SECONDARY OUTCOMES:
The Functional Independence Measure for Children (WeeFIM): | 8 weeks
  WeeFIM is an 18-item, 7-level ordinal scale instrument that measures a child's consistent performance in essential daily functional skills. The method measures functional performance in three domains: self-care, mobility, and cognition. The lowest total score is 18 and the highest total score 126.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Hayatabad Medical Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters C, Chang A, Morales A, Barnes K, Allegretti A. An integrative review of assessments used in occupational therapy interventions for children with cerebral palsy. Brazilian J Occup Ther. 2019;27(1):168-85.
- [Background] Klingels K, De Cock P, Molenaers G, Desloovere K, Huenaerts C, Jaspers E, Feys H. Upper limb motor and sensory impairments in children with hemiplegic cerebral palsy. Can they be measured reliably? Disabil Rehabil. 2010;32(5):409-16. doi: 10.3109/09638280903171469. PMID 20095955
- [Background] Kassee C, Hunt C, Holmes MWR, Lloyd M. Home-based Nintendo Wii training to improve upper-limb function in children ages 7 to 12 with spastic hemiplegic cerebral palsy. J Pediatr Rehabil Med. 2017 May 17;10(2):145-154. doi: 10.3233/PRM-170439. PMID 28582885
- [Background] Camerota F, Galli M, Cimolin V, Celletti C, Ancillao A, Blow D, Albertini G. Neuromuscular taping for the upper limb in Cerebral Palsy: A case study in a patient with hemiplegia. Dev Neurorehabil. 2014 Dec;17(6):384-7. doi: 10.3109/17518423.2013.830152. Epub 2013 Oct 2. PMID 24087981
- [Background] Wang TN, Liang KJ, Liu YC, Shieh JY, Chen HL. Psychometric and Clinimetric Properties of the Melbourne Assessment 2 in Children With Cerebral Palsy. Arch Phys Med Rehabil. 2017 Sep;98(9):1836-1841. doi: 10.1016/j.apmr.2017.01.024. Epub 2017 Feb 28. PMID 28254639